CLINICAL TRIAL: NCT02532634
Title: Comparison of Ramosetron, Aprepitant, and Dexamethasone (RAD) With Palonosetron, Aprepitant, and Dexamethasone (PAD) for Prevention of Nausea and Vomiting Induced by Highly Emetogenic Chemotherapy
Brief Title: Ramosetron, Aprepitant, and Dexamethasone Versus Palonosetron, Aprepitant, and Dexamethasone
Acronym: RAPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kangdong Sacred Heart Hospital (Other)
Collaborators: The Catholic University of Korea (Other); Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Principal Investigator, Kwon, Jung Hye, Associate Professor, Kangdong Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KJH-2015-01
Record Dates: First submitted 2015-08-23; First posted 2015-08-26 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Cancer; Tumors
Keywords: ramosetron; palonosetron; chemotherapy induced nausea and vomiting
MeSH Terms: conditions — Neoplasms; Vomiting | interventions — ramosetron; Aprepitant; Dexamethasone; Palonosetron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ramosetron, aprepitant, dexamethasone (Experimental): 1. Ramosetron 0.3mg IV day1
  2. Aprepitant 125mg PO qd day1, 80mg po qd day 2, 3
  3. Dexamethasone 12mg IV or PO qd day1, 8mg PO day 2, 3, 4
  Interventions: Drug: ramosetron, aprepitant, dexamethasone
- palonosetron, aprepitant, dexamethasone (Active Comparator): 1. Palonosetron 0.25mg IV day1
  2. Aprepitant 125mg PO qd day1, 80mg po qd day 2, 3
  3. Dexamethasone 12mg IV or PO qd day1, 8mg PO day 2, 3, 4
  Interventions: Drug: palonosetron, aprepitant, dexamethasone

INTERVENTIONS:
Drug: ramosetron, aprepitant, dexamethasone — ramosetron 0.3 mg IV D1 aprepitant 125 mg PO D1, 80 mg PO D2, 80 mg PO D3 dexamethasone 12 mg PO D1, 8 mg PO D2-4
  Other Names: ramosetron(nasea); aprepitant(emend)
  Arms: ramosetron, aprepitant, dexamethasone
Drug: palonosetron, aprepitant, dexamethasone — palonosetron 0.25 mg IV D1 aprepitant 125 mg PO D1, 80 mg PO D2, 80 mg PO D3 dexamethasone 12 mg PO D1, 8 mg PO D2-4
  Other Names: palonosetron(aloxi); aprepitant(emend)
  Arms: palonosetron, aprepitant, dexamethasone

SUMMARY:
The purpose of this study is to compare the anti-emetic effect of ramosetron plus aprepitant and dexamethasone with palonosetron plus aprepitant and dexamethasone in patients receiving highly emetogenic chemotherapy.

DETAILED DESCRIPTION:
Currently, palonosetron is the clinically preferred antiemetic for Chemotherapy-induced nausea and vomiting (CINV).However the best 5-hydroxytryptamine 3 receptor (5-HT3R) antagonists for use in a triple drug combination for high emetogenic chemotherapy(HEC) has not yet been determined in randomized trials. Previous anti-emetic guidelines stated that the anti-emetic activities of 5-HT3R antagonists were similar at equivalent doses. Based on the meta-analysis of various 5-HT3R antagonists in double regimens, the NCCN guideline has suggested palonosetron as a preferred 5-HT3R antagonist in the triple antiemetic drug combination. But in Asia, RAD is one of the most popular treatments for HEC-treated cancer patients. However, the lack of clinical studies has precluded the recommendation of RAD as a standard regimen for HEC-induced CINV. In two previous studies conducted in Korea, RAD regimen showed significant efficacy for prevention of CINV which is comparable to the efficacy reported from the studies evaluating with PAD regimen. If the efficacy of RAD regimen is evidently proven by this kind of randomized multicenter-trial, RAD regimen can be more recommended as a standard regimen for HEC-induced CINV.

ELIGIBILITY:
Inclusion Criteria:

* The patient's age is ≥ 19 years old
* Histologically or cytologically confirmed solid tumor
* Patients diagnosed as malignancy who will be treated with highly emetogenic chemotherapeutic agents (NCCN guideline v2.0, 2014 anti-emesis). (Cisplatin dosage is over 50mg/m2, combination therapy is available with other chemotherapeutic agents and including lymphoma)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Available oral administration of study drugs
* Adequate organ functions as follows: 1) Hematologic - white blood cell count (WBC) ≥ 3000 microliter (microL) or Neutrophil≥ 1500 micro/L, Platelet ≥ 100,000/microL; 2) Serum Creatinine ≤ 1.5 times upper limit of normal; 3) Hepatic function - Total bilirubin, AST, ALT ≤2.5 times upper limit of normal, ALP ≤ 2 times upper limit of normal( except ALP increasing due to bone metastasis
* Patients with normal range of serum K, Mg and hold serum Ca over lower limit of normal range
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital

Exclusion Criteria:

* Patients with severe Hypertension, severe Heart disease, congenital long QT syndrome, bradyarrhythmia severe kidney disease(serum creatinine≥3㎎/㎗), liver disease (AST, ALT ≥ 2.5 times of upper normal range, ALP ≥ 2 times of upper normal range)
* Patients with GI obstruction, active gastric ulcer or other diseases that could provoke nausea and vomiting
* Patients who have nausea and vomiting within 1 week before chemotherapy
* Patients who should take steroid, antiemetics, antipsychotic agent including benzodiazepine, pimozide, terfenadine, astemizole, cisapride, rifampin, carbamazepine, phenytoin, ketoconazole, itraconazole, nefazodone, troleandomycin, clarithromycin, ritonavir or nelfinavir, selective serotonin reuptake inhibitors, serotonin-norepinephrine reuptake inhibitors for the treatment of other diseases
* Patients with brain tumor, brain metastasis or seizure
* Patients receiving chemotherapy within 6 months before enrollment
* Patients who need radiation therapy during study period or receiving radiation therapy within 2 weeks before chemotherapy
* Patients who have known allergy or severe side effect on study drugs(5-HT3 antagonist and aprepitant)
* Pregnant or lactating women, or women who wish to become pregnant
* Patients with drug abuse, a mental disease and difficult to communicate with investigators
* Others whom the investigator judges inappropriate as subjects for this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2018-05-08 (Actual)

PRIMARY OUTCOMES:
To compare the overall complete response (CR) of RAD to PAD (Overall CR defined as no emesis, no rescue medication, at cycle 1 | 0-120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Hyoung Kang, Ph.D, Principal Investigator — The Catholic University of Korea; Jung Hye Kwon, PhD, Study Director — Kangdong Sacred Heart Hospital
Locations (10):
- South Korea (10):
  - St. Vincent'S Hospital, Suwon, Gyeonggi-do
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospita, Daejeon
  - Pusan National University Hospital, Pusan
  - Kangbuk Samsung Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Severance Hospital, Seoul
  - Ajou University Hospital, Suwon